CLINICAL TRIAL: NCT03933501
Title: The Use of Amoxicillin and Metronidazole in Association With Non-surgical Therapy in Aggressive Periodontitis Treatment
Brief Title: Amoxicillin and Metronidazole in Association With Non-surgical Therapy in Aggressive Periodontitis Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Renato Casarin, Professor at Piracicaba Dental School, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06/0024
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Generalized Aggressive Periodontitis
Keywords: Aggressive periodontitis; anti-infective agents; debridement; randomized clinical trial; ultrasonic
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Amoxicillin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- FMUD + AM (Experimental): One session of full-mouth ultrasonic debridement (FMUD) with a time limit of 45 minutes plus 375 mg amoxicillin and 250 mg metronidazole (AM) prescribed on the day of treatment, every 8 hours for 7 days.
  Interventions: Drug: amoxicillin and metronidazole
- FMUD (Placebo Comparator): One session of full-mouth ultrasonic debridement (FMUD) with a time limit of 45 minutes plus two distinct placebo pills prescribed on the day of treatment and taken every 8 hours for 7 days.
  Interventions: Drug: Placebos
- SRP + AM (Experimental): Four sessions (1/week) of scaling and root planning, plus 375 mg amoxicillin and 250 mg metronidazole (AM) prescribed on the last session of treatment and taken every 8 hours for 7 days.
  Interventions: Drug: amoxicillin and metronidazole
- SRP (Placebo Comparator): Four sessions (1/week) of scaling and root planning, plus two distinct placebo pills prescribed on the last session of treatment and taken every 8 hours for 7 days.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: amoxicillin and metronidazole — 375 mg amoxicillin and 250 mg metronidazole prescribed on the day of treatment, every 8 hours for 7 days.
  Arms: FMUD + AM; SRP + AM
Drug: Placebos — Two distinct placebo pills prescribed on the day of treatment and taken every 8 hours for 7 days.
  Arms: FMUD; SRP

SUMMARY:
This study is designed as a parallel, masked, randomized, placebo-controlled clinical trial to assess the clinical, microbiological, and immunological outcomes of scaling and root planning (SRP) or full-mouth ultrasonic debridement (FMUD) with AM (Amoxicillin + Metronidazole) for the treatment of Generalized Aggressive Periodontitis (GAgP).

DETAILED DESCRIPTION:
Forty eight GAgP patients were divided into 4 groups: the SRP group (n = 12), which received SRP plus placebo, and the SRP+AM group (n = 12), which received SRP and 375mg amoxicillin plus 250 mg metronidazole for 7 days, the FMUD group (n = 12), which received FMUD plus placebo, and the FMUD+AM group (n = 12), which received FMUD and 375mg amoxicillin plus 250 mg metronidazole for 7 days. The following clinical outcomes were tested: plaque and bleeding on probing indices, pocket probing depth (PD), relative gingival margin position (GMP), and relative clinical attachment level (CAL). The total amount of Porphyromonas gingivalis (Pg), Aggregatibacter actinomycetemcomitans (Aa), Tannerella forsythia (Tf), and gingival crevicular fluid (GCF) concentration of interleukin (IL)-10 and IL-1b were also determined. All clinical, microbiological, and immunological parameters were assessed at baseline and at 3 and 6 months post-therapy. The ANOVA/Tukey test was used for statistical analysis (a = 5%).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of GAgP;
* presence of 20 teeth;
* presence of teeth presenting PD>5 mm with bleeding on probing (BOP) and 2 teeth with PD>7mm (including incisors and first molars, in addition to two other non-contiguous teeth between them);
* good general health;
* <35 years of age.

Exclusion Criteria:

* were pregnant or lactating;
* were suffering from any other systemic diseases (e.g., cardiovascular, diabetes);
* received antimicrobials in the previous 3 months;
* were taking long-term anti-inflammatory drugs;
* received a course of periodontal treatment within the last 6 months;
* smoked

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2008-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change of the baseline relative clinical attachment level at 6 months | Baseline, 3 months and 6 months
  distance from the bottom of the pocket to the stent margin.

SECONDARY OUTCOMES:
Change of the baseline probing depth at 6 months | Baseline, 3 months and 6 months
  Distance from the bottom of pocket to gingival margin;
Change of the baseline inflammatory markers levels in gingival crevicular fluid (pg/uL) at 6 months | Baseline, 3 months and 6 months
  Concentration of IL-1β, IL-10 released in gingival crevicular fluid
Change in the microbial composition at 6 months | Baseline, 3 months and 6 months
  Concentration of bacteria in the subgingival biofilm

REFERENCES:
- [Derived] Taiete T, Monteiro MF, Casati MZ, do Vale HF, Ambosano GMB, Nociti FH, Sallum EA, Casarin RCV. Local IL-10 level as a predictive factor in generalized aggressive periodontitis treatment response. Scand J Immunol. 2019 Dec;90(6):e12816. doi: 10.1111/sji.12816. Epub 2019 Oct 3. PMID 31448837